CLINICAL TRIAL: NCT04113252
Title: The Economy of Pain: A Pilot Study of the Impact of an Opioid Buyback Program
Brief Title: Impact of Coaching Patients on Pain Control With and Without Financial Incentivization
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Too difficult to see patients in required time intervals.
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB00058073
Record Dates: First submitted 2019-10-01; First posted 2019-10-02 (Actual); Last update posted 2022-05-12 (Actual); Status verified 2021-08

CONDITIONS: Opioid Use
Keywords: opioid buyback; opioid misuse prevention

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1--Diary and Possible Opioid Return Incentive (Experimental): Participants in this arm will be given incentives upon return of completed diary and will have the possibility to earn incentives for returning any leftover tablets to the study team.
  Interventions: Other: Possible Incentive for Tablet Return; Other: Incentive for Completed Diary
- Group 2--Diary, Coaching, Possible Opioid Return Incentive (Experimental): Participants in this arm will be given coaching. They will also be given incentives upon return of completed diary and will have the possibility to earn incentives for returning any leftover tablets to the study team.
  Interventions: Other: Possible Incentive for Tablet Return; Other: Incentive for Completed Diary; Behavioral: Coaching
- Group 3--Diary and coaching (Experimental): Participants in this arm will be given coaching. They will also be given incentives upon return of completed diary.
  Interventions: Other: Incentive for Completed Diary; Behavioral: Coaching

INTERVENTIONS:
Other: Possible Incentive for Tablet Return — Subjects who return completed diary will have the possibility to receive money for returned opioid tablets.
  Arms: Group 1--Diary and Possible Opioid Return Incentive; Group 2--Diary, Coaching, Possible Opioid Return Incentive
Other: Incentive for Completed Diary — Subjects who return completed diary will receive a gift card.
Behavioral: Coaching — Subjects will receive coaching prior to starting pain medication.
  Arms: Group 2--Diary, Coaching, Possible Opioid Return Incentive; Group 3--Diary and coaching

SUMMARY:
Opioids are commonly prescribed pain medications, but they can lead to addiction. The study team is trying to determine if providing someone with an incentive (money in the form of a Visa gift card) to use less pain medications will result in study participants actually using fewer pain tablets than allowed by their health care provider. The study team also wants to know if providing the incentive (the Visa gift card alone) works the same as the incentive (the Visa gift card) plus providing additional information about addiction and alternative pain management.

DETAILED DESCRIPTION:
Study participants will receive the standard of care for pain management at discharge. If study participants were not hospitalized at discharge, the study team will begin that standard of pain management at the participant's first outpatient clinic visit. Study participants will be randomized to 1 of 3 groups. All groups will receive a gift card if participants return the completed medication diary to the study team.

* Group 1 will complete a medication diary. Also, group 1 will be encouraged to return any unused tablets to the study clinic.
* Group 2 will be asked to complete a medication diary. Group 2 will also have a 50/50 chance of receiving money for each unused opioid tablet returned to the study clinic.
* Group 3 will be the same as group 2 except in addition, they will be given a coaching session about the use of pain medication and a simple way that may help participants use less opioid pain medication.

ELIGIBILITY:
Inclusion Criteria:

* Patients suffering from a burn injury of one or both hands/upper extremities
* Patients staying less than 2 midnights after date of injury or presenting for first visit to the clinic 4 or less days after injury
* Patients able to self-administer their oxycodone.
* Aged 18-89 years old

Exclusion Criteria:

* No burns on either hand or upper extremity
* Patients suffering chemical or electrical burns
* Patients with other traumatic injuries for which they might require opioids/pain treatment
* Patients taking opioids prior to injury
* Patients who are discharged with prescriptions other than oxycodone with a dosage of 5 milligrams by mouth every six hours as needed

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-05 (Estimated); Primary Completion 2022-08 (Estimated); Study Completion 2022-08 (Estimated)

PRIMARY OUTCOMES:
Mean number of opioid tablets used daily | up through two weeks

CONTACTS AND LOCATIONS:
Overall Officials: John K Bailey, MD, Principal Investigator — Wake Forest University Health Sciences

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF